CLINICAL TRIAL: NCT02798159
Title: A Randomized, Placebo Control, Double-blinded, Double-dummy, Phase 2/3 Combination Study to Evaluate the Safety and Efficacy of TD0025 (Rocket1h) Compared With Sildenafil Citrate for Treatment of Erectile Dysfunction
Brief Title: Safety and Efficacy of TD0025 (Rocket1h) for Treatment of Erectile Dysfunction
Acronym: TD0025
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vietstar Biomedical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TD0025
Record Dates: First submitted 2016-06-04; First posted 2016-06-14 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2016-06

CONDITIONS: Erectile Dysfunction
Keywords: Sexual Dysfunction; Physiological Sexual Dysfunctions; Psychological Sexual and Gender Disorders; Sildenafil
MeSH Terms: conditions — Erectile Dysfunction; Sexual Dysfunction, Physiological | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part A- Arm 1 (Experimental): Investigational dose = 0.25 time of the expected dose. The drug should not be taken more than one time a day or 3 times a week Drug: TD0025 Administered orally once a day, 5 hours before sexual activity, for 1 month.
  Interventions: Drug: TD0025
- Part A- Arm 2 (Experimental): Investigational dose = 0.5 time of the expected dose. The drug should not be taken more than one time a day or 3 times a week Drug: TD0025 Administered orally once a day, 5 hours before sexual activity, for 1 month.
  Interventions: Drug: TD0025
- Part A- Arm 3 (Experimental): Investigational dose = 1 time of the expected dose. The drug should not be taken more than one time a day or 3 times a week Drug: TD0025 Administered orally once a day, 5 hours before sexual activity, for 1 month.
  Interventions: Drug: TD0025
- Part A- Arm 4 (Experimental): Investigational dose = 1.25 time of the expected dose. The drug should not be taken more than one time a day or 3 times a week Drug: TD0025 Administered orally once a day, 5 hours before sexual activity, for 1 month.
  Interventions: Drug: TD0025
- Part B- Arm 1 (Experimental): Investigational dose = optimal dose in Part A. The drug should not be taken more than one time a day or 3 times a week.
  Drug: TD0025 Administered orally once a day, 5 hours before sexual activity, for 1 month
  Interventions: Drug: TD0025
- Part B- Arm 2 (Active Comparator): Sildenafil Citrate 50 mg on demand The drug should not be taken more than one time a day or 3 times a week. Administered orally once a day, 1 hour before sexual activity, for 1 month
  Interventions: Drug: Sildenafil Citrate 50mg

INTERVENTIONS:
Drug: TD0025
  Arms: Part A- Arm 1; Part A- Arm 2; Part A- Arm 3; Part A- Arm 4; Part B- Arm 1
Drug: Sildenafil Citrate 50mg
  Arms: Part B- Arm 2

SUMMARY:
The purpose of this study is to identify the optimal dose(s) of TD0025 for treatment of erectile dysfunction (phase II) and to investigate if treatment of erectile dysfunction with the optimal dose of TD0025 taken as needed over one month is non-inferior than Sildenafil Citrate taken as needed over one month (phase III)

ELIGIBILITY:
Main Inclusion Criteria:

* History of Erectile Dysfunction (ED) of at least 1 month duration.
* Anticipate having the same adult female sexual partner during the study.
* Agree not to use any other treatment for ED and to participate in recording responses to questionnaires and other instruments used in this study.
* Sign the informed consent form

Main Exclusion Criteria:

* ED caused by other primary sexual disorders, history of radical prostatectomy or other pelvic surgery with subsequent failure to achieve any erection, or history of penile implant or clinically significant penile deformity
* ED caused by untreated or inadequately treated endocrine disease
* Current treatment with doxazocin, nitrates, cancer chemotherapy, or anti-androgens
* Severe renal or hepatic impairment, history of malignant hypertension
* Presence or history of specific heart conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
PART A- PHASE II: Change From Baseline to 4 Weeks of the International Index of Erectile Function (IIEF), question # 3 and #4 | Baseline, 4 weeks
PART B- PHASE III: Change From Baseline to 4 Weeks of the International Index of Erectile Function (IIEF) Erectile Function (EF) Domain | Baseline, 4 weeks

SECONDARY OUTCOMES:
PART A- PHASE II: Change From Baseline to 4 Weeks of the International Index of Erectile Function (IIEF), Erectile Function (EF) Domain | Baseline, 4 weeks
PART A- PHASE II: Change From Baseline to 4 Weeks of the International Index of Erectile Function (IIEF), Orgasmic Function Domain | Baseline, 4 weeks
PART A- PHASE II: Change From Baseline to 4 Weeks of the International Index of Erectile Function (IIEF), Sexual Desire Domain | Baseline, 4 weeks
PART A- PHASE II: Change From Baseline to 4 Weeks of the International Index of Erectile Function (IIEF), Intercourse Satisfaction Domain | Baseline, 4 weeks
PART A- PHASE II: Change From Baseline to 4 Weeks of the International Index of Erectile Function (IIEF), Overall Satisfaction Domain | Baseline, 4 weeks
PART A- PHASE II: The percentage of patients with abnormal Testosterone, FSH, LH and Androgen Serum Levels at Baseline and after 4 weeks of treatment | Baseline, 4 weeks
PART A- PHASE II: The percentage of patients with abnormal hematology and biochemistry laboratory values at baseline and after 4 weeks of treatment | Baseline, 4 weeks
PART B- PHASE III: Change From Baseline to 4 Weeks of the International Index of Erectile Function (IIEF), Orgasmic Function Domain | Baseline, 4 weeks
PART B- PHASE III: Change From Baseline to 4 Weeks of the International Index of Erectile Function (IIEF), Sexual Desire Domain | Baseline, 4 weeks
PART B- PHASE III: Change From Baseline to 4 Weeks of the International Index of Erectile Function (IIEF), Intercourse Satisfaction Domain | Baseline, 4 weeks
PART B- PHASE III: Change From Baseline to 4 Weeks of the International Index of Erectile Function (IIEF), Overall Satisfaction Domain | Baseline, 4 weeks
PART B- PHASE III: Time to Discontinuation of Randomized Treatment | Baseline up to 30 days
PART B- PHASE III: Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) Questionnaire at 4 Weeks | 4 weeks
PART B- PHASE III: Change From Baseline to 4 Weeks of the Sexual Relationship Domain of the Self-Esteem and Relationship (SEAR) Questionnaire | Baseline, 4 weeks
PART B- PHASE III: Change From Baseline to 4 Weeks of the Confidence Domain of the Self-Esteem and Relationship (SEAR) Questionnaire | Baseline, 4 weeks
PART B- PHASE III: Change From Baseline to 4 Weeks of the Self Esteem Domain of the Self-Esteem and Relationship (SEAR) Questionnaire | Baseline, 4 weeks
PART B- PHASE III: Change From Baseline to 4 Weeks of the Overall Relationship Domain of the Self-Esteem and Relationship (SEAR) Questionnaire | Baseline, 4 weeks
PART B- PHASE III: The percentage of patients with abnormal Testosterone, FSH, LH and Androgen Serum Levels at Baseline and after 4 weeks of treatment | Baseline, 4 weeks
PART B- PHASE III: The percentage of patients with abnormal hematology and biochemistry laboratory values at baseline and after 4 weeks of treatment | Baseline, 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nguyen Quang, MD. PhD., Principal Investigator — Men Sexual Health Centre, Vietnam- Germany Hospital
Locations (1):
- Men Sexual Health Centre; Vietnam- Germany Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided